CLINICAL TRIAL: NCT01220271
Title: Phase 1b/2a Study Combining LY2157299 With Standard Temozolomide-based Radiochemotherapy in Patients With Newly Diagnosed Malignant Glioma
Brief Title: A Study Combining LY2157299 With Temozolomide-based Radiochemotherapy in Patients With Newly Diagnosed Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11585; H9H-MC-JBAI (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Glioma
Keywords: Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — LY-2157299; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1: 160 mg LY2157299 (Experimental): During Radiation therapy:
  * Radiation:Approximate 1.8 - 2.0 Gy x 30 fractions. Approximate total dose = 60.0 Gy taken 5 days per week for 6 weeks.
  * LY2157299: 80 mg taken twice daily for 14 days on followed 14 days of pause. This on/off schedule constitutes a cycle of 28 days.
  * Temozolomide: 75 mg/m2 taken daily for 6 weeks.
  After Radiation Therapy:
  * LY2157299: 80 mg taken twice daily for 14 days on followed 14 days of pause. This on/off schedule constitutes a cycle of 28 days. Taken for a 6 cycles.
  * Temozolomide: 150 mg/m2 and then 200 mg/m2 daily during the off time of LY2157299. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  Interventions: Drug: LY2157299; Drug: Radiation; Drug: Temozolomide
- Phase 1: 300 mg LY2157299 (Experimental): During Radiation therapy:
  * Radiation:Approximate 1.8 - 2.0 Gy x 30 fractions. Approximate total dose = 60.0 Gy taken 5 days per week for 6 weeks.
  * LY2157299: 150 mg taken twice daily for 14 days on followed 14 days of pause. This on/off schedule constitutes a cycle of 28 days.
  * Temozolomide: 75 mg/m2 taken daily for 6 weeks.
  After Radiation Therapy:
  * LY2157299: 150 mg taken twice daily for 14 days on followed 14 days of pause. This on/off schedule constitutes a cycle of 28 days. Taken for a 6 cycles.
  * Temozolomide: 150 mg/m2 and then 200 mg/m2 daily during the off time of LY2157299. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  Interventions: Drug: LY2157299; Drug: Radiation; Drug: Temozolomide
- Phase 2: Established dose LY2157299 (Experimental): During Radiation therapy:
  * Radiation:Approximate 1.8 - 2.0 Gy x 30 fractions. Approximate total dose = 60.0 Gy taken 5 days per week for 6 weeks.
  * LY2157299: Phase 1 established dose taken twice daily for 14 days on followed 14 days of pause. This on/off schedule constitutes a cycle of 28 days.
  * Temozolomide: 75 mg/m2 taken daily for 6 weeks.
  After Radiation Therapy:
  * LY2157299: Phase 1 established dose taken twice daily for 14 days on followed 14 days of pause. This on/off schedule constitutes a cycle of 28 days. Taken for a 6 cycles.
  * Temozolomide: 150 mg/m2 and then 200 mg/m2 daily during the off time of LY2157299. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  Interventions: Drug: LY2157299; Drug: Radiation; Drug: Temozolomide
- Phase 2: no LY2157299 (control) (Experimental): During Radiation therapy:
  * Radiation:Approximate 1.8 - 2.0 Gy x 30 fractions. Approximate total dose = 60.0 Gy taken 5 days per week for 6 weeks.
  * Temozolomide: 75 mg/m2 taken daily for 6 weeks.
  After Radiation Therapy:
  Temozolomide: 150 mg/m2 and then 200 mg/m2 daily during the off time of LY2157299. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  Interventions: Drug: Radiation; Drug: Temozolomide

INTERVENTIONS:
Drug: LY2157299 — Administered orally
  Arms: Phase 1: 160 mg LY2157299; Phase 1: 300 mg LY2157299; Phase 2: Established dose LY2157299
Drug: Radiation — Administered as approved
Drug: Temozolomide — Administered orally

SUMMARY:
The purpose of this trial is to show proof of concept that by blocking the Transforming Growth Factor-beta signaling pathway in patients with Glioblastoma, there will be clinical benefit.

Phase 1b: To determine the safe and tolerable dose of LY2157299 in combination with radiochemotherapy with temozolomide for Phase 2 in patients with glioma eligible to receive radiochemotherapy with temozolomide (e.g. newly diagnosed malignant glioma World Health Organization Grade III and IV).

Phase 2a: To confirm the tolerability and evaluate the pharmacodynamic effect of LY2157299 in combination with standard radiochemotherapy in patients with newly diagnosed glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven, newly diagnosed and untreated intracranial glioblastoma including lower grade glioma which evolved into glioblastoma and who have not received any radiochemotherapy or who have World Health Organization Grade III malignant glioma (e.g., Anaplastic Astrocytomas, Anaplastic Oligoastrocytomas, Anaplastic Oligodendroglioma) (Phase 1b only) will be eligible for this protocol
* Biopsy or resection must have been performed no more than 6 weeks prior to treatment
* An Magnetic Resonance Imaging must be obtained within 72 hours after surgery, preferably within 48 hours
* Patient must not have had prior cranial radiation therapy
* Patients must not have received prior cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy for brain tumors Patients who received Gliadel wafers at the time of original resection will be excluded
* Patients must plan to begin partial brain radiotherapy within 2-6 weeks after surgery. Regular fractionated radiotherapy with photons (in any planning mode and possibly image-guided or stereotactic if deemed necessary) is performed according to the discretion of the investigator
* Patients must be willing to forego other cytotoxic and noncytotoxic drug therapy against the tumor while being treated with LY2157299 and temozolomide
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study
* Patients must have performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Patients must have adequate hematologic, hepatic and renal function
* Male and female patients with reproductive potential must use an approved contraceptive method,during and for 6 months after discontinuation of study treatment Women of childbearing potential must have a negative human chorionic gonadotropin pregnancy test documented within 14 days prior to treatment

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or not approved use of a drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have moderate or severe cardiac disease as defined by any of the following:

  * Have the presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension
  * Have documented major electrocardiogram (ECG) abnormalities that are symptomatic and are not medically controlled
  * Have major abnormalities documented by echocardiography with Doppler
  * Have predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress
* Are unable to swallow tablets or capsules
* Are pregnant or breastfeeding
* Have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and stopped all therapy for that disease for a minimum of 3 years are ineligible
* Have active infection that would interfere with the study objectives or influence the study compliance
* Stereotactic radiosurgery, such as Gamma-Knife treatment, and brachytherapy are not allowed in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-04; Primary Completion 2015-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Phase 1: Recommended dose for Phase 2 portion | Baseline to phase 1 completion
Phase 2: Relationship of change in response biomarker to clinical benefit | Baseline through discontinuation from any cause

SECONDARY OUTCOMES:
Phase 1: Pharmacokinetics - Concentration Maximum | Baseline, prior to first dose of cycle 1 and 2 and on days 1, 3, 8, 14, 15 and 16
Phase 1: Number of patients with a tumor response | Baseline to Progressive Disease
Phase 2: Overall Survival at 12 Months | Randomization to date of death from any cause at 12 months
Phase 2: Overall Survival | Randomization to date of death from any cause
Phase 2: Progression Free Survival | Randomization to measured progressive disease or death from any cause
Phase 2: Proportion of patients achieving an objective response (Response Rate) | Randomization to measured progressive disease
Phase 2: Duration of tumor Response | Time of response to measured progressive disease or death from any cause
Phase 2: Time to Treatment Failure | Randomization to the date of discontinuation of study treatment due to adverse event, progression of disease, or death from any cause
Phase 1: Pharmacokinetics - Time to Concentration Maximum | Baseline, prior to first dose of cycle 1 and 2 and on days 1, 3, 8, 14, 15 and 16
Phase 1: Pharmacokinetics - Area under the Curve | Days 12 to 14 in cycle 1 and in cycle 3
Phase 2: Change from baseline in MD Anderson Symptom Inventory - Brain Tumor | Baseline, 30 day post study day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid

REFERENCES:
- [Derived] Wick A, Desjardins A, Suarez C, Forsyth P, Gueorguieva I, Burkholder T, Cleverly AL, Estrem ST, Wang S, Lahn MM, Guba SC, Capper D, Rodon J. Phase 1b/2a study of galunisertib, a small molecule inhibitor of transforming growth factor-beta receptor I, in combination with standard temozolomide-based radiochemotherapy in patients with newly diagnosed malignant glioma. Invest New Drugs. 2020 Oct;38(5):1570-1579. doi: 10.1007/s10637-020-00910-9. Epub 2020 Mar 5. PMID 32140889